CLINICAL TRIAL: NCT03125356
Title: Low-calorie Sweeteners and Adipose Signaling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 111635
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Nutritional and Metabolic Diseases
Keywords: diet soda; low-calorie sweeteners; obesity
MeSH Terms: conditions — Nutritional and Metabolic Diseases; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diet Soda (Experimental): Subjects will be asked to consume a diet soda three times daily for eight weeks.
  Interventions: Other: Diet Soda

INTERVENTIONS:
Other: Diet Soda — Subjects will be asked to consume diet soda three times daily for eight weeks.

SUMMARY:
The purpose of this study is to determine whether eight weeks of low-calorie sweetener (LCS) exposure exerts cardiovascular and/or metabolic effects among LCS-naïve overweight and obese adolescents and young adults. We will examine changes in gene expression in subcutaneous fat and will correlate these molecular changes with plasma biochemistry.

DETAILED DESCRIPTION:
The proposed study will investigate LCS-induced changes in metabolically "at-risk" young adults, under conditions that reflect typical beverage consumption. We will first identify molecular pathways potentially affected by LCS (adipose transcriptomics via global RNAseq) and then identify links between LCS-induced gene expression changes and circulating levels of key metabolic biomarkers and clinical outcomes. We will perform subcutaneous adipose biopsies before and after consumption of 12 ounces of diet soda three times daily for eight weeks. Within-subjects changes in adipose gene expression will be evaluated using RNAseq. We will then correlate transcriptomic changes with circulating levels of key inflammatory and metabolic biomarkers, to provide mechanistic insight into which pathways drive clinically-relevant LCS-induced metabolic impairments. We will measure glucose, insulin, inflammatory markers and adipose-derived hormones before and after eight weeks of LCS exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. 18-25 years of age
3. Overweight and mild to moderate obesity (25 ≤ body mass index (BMI) <35 kg/m2)
4. Consumption of <1 food/beverage with sucralose and/or acesulfame-potassium per month
5. Able and willing to comply with all study procedures for the duration of the study

Exclusion Criteria:

1. Overt diabetes
2. Renal/gastrointestinal conditions
3. Pregnant/lactating
4. Recent significant weight change
5. Acute illness (w/fever)
6. Antibiotics in past 3 months
7. Use of illegal drugs/condition limiting ability to give consent.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Transcriptomics | Pre/post 8 weeks of diet soda
  Within-subjects changes in adipose gene expression will be evaluated using RNAseq

CONTACTS AND LOCATIONS:
Locations (1):
- Milken Institute School of Public Health and GW Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sylvetsky AC, Clement RA, Stearrett N, Issa NT, Dore FJ, Mazumder R, King CH, Hubal MJ, Walter PJ, Cai H, Sen S, Rother KI, Crandall KA. Consumption of sucralose- and acesulfame-potassium-containing diet soda alters the relative abundance of microbial taxa at the species level: findings of two pilot studies. Appl Physiol Nutr Metab. 2024 Jan 1;49(1):125-134. doi: 10.1139/apnm-2022-0471. Epub 2023 Oct 30. PMID 37902107